CLINICAL TRIAL: NCT02716948
Title: A Pilot Study of Stereotactic Radiosurgery Combined With Nivolumab in Patients With Newly Diagnosed Melanoma Metastases in the Brain and Spine
Brief Title: SRS and Nivolumab in Treating Patients With Newly Diagnosed Melanoma Metastases in the Brain or Spine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Accuray Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J15214; NCI-2016-00370 (Registry Identifier: CTRP); IRB00086553 (Other: JHMIRB)
Record Dates: First submitted 2016-03-17; First posted 2016-03-23 (Estimated); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Metastatic Malignant Neoplasm in the Brain; Metastatic Malignant Neoplasm in the Spine; Stage IV Skin Melanoma
MeSH Terms: conditions — Brain Neoplasms; Melanoma | interventions — Nivolumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (nivolumab, stereotactic radiosurgery) (Experimental): Patients receive nivolumab IV over 60 minutes on day 1. Patients then undergo stereotactic radiosurgery on day 8 per standard of care. Courses with nivolumab repeats every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; ONO-4538; Opdivo
Radiation: Stereotactic Radiosurgery — Undergo stereotactic radiosurgery
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; Stereotactic Radiation Therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery

SUMMARY:
This phase I pilot trial studies the side effects of stereotactic radiosurgery and nivolumab in treating patients with newly diagnosed melanoma that has spread to the brain or spine. Stereotactic radiosurgery is a specialized radiation therapy that delivers a single, high dose of radiation directly to the tumor to more precisely target the cancer. Monoclonal antibodies, such as nivolumab may interfere with the ability of tumor cells to grow and spread. Giving stereotactic radiosurgery together with nivolumab may be a better treatment for melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety profile of stereotactic radiosurgery with nivolumab in combination to treat patients with newly diagnosed melanoma brain or spinal metastases.

SECONDARY OBJECTIVES:

I. To estimate local control rate in brain and spine. II. To estimate systematic control rate. III. To estimate progression-free survival.

TERTIARY OBJECTIVES:

I. To explore peripheral blood immune response during and after treatment.

OUTLINE:

Patients receive nivolumab intravenously (IV) over 60 minutes on day 1. Patients then undergo stereotactic radiosurgery on day 8 per standard of care. Courses with nivolumab repeats every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 10 weeks, and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of melanoma; the pathologic confirmation may be from another metastatic site or from metastatic brain or spine lesions
* Patients must have stage IV melanoma, with newly identified brain or spine metastases
* Patients must have measurable lesion in the brain or spine that is >= 3 mm seen on magnetic resonance imaging (MRI) with contrast; NOTE: contrasted pre-treatment MRI scan must be obtained =< 21 days prior to stereotactic radiosurgery treatment
* Karnofsky performance scale >= 70%
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 2 x institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/ alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR according to Johns Hopkins MRI policy
* Women of child bearing potential (WOCBP) must use a reliable form of contraception during the study treatment period and for up to 12 weeks following the last dose of study drug
* Men must agree to the use of male contraception during the study treatment period and for at least 12 weeks after the last dose of study drug
* Ability to understand and the willingness to sign written informed consent document(s)

Exclusion Criteria:

* Prior whole brain radiation or conventional radiation to the spine at the site of new lesion
* Prior chemotherapy within 28 days of starting treatment
* Prior therapy with investigational drugs within 28 days or at least 5 half-lives (whichever is longer) before study administration
* Prior therapy with an anti- programmed cell death 1 (PD-1), anti- programmed cell death-ligand 1 (PD-L1), or anti-PDL-2 antibody
* Neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Known allergy to compounds of similar chemical or biologic composition to nivolumab
* Pregnant or breastfeeding women
* Known history of human immunodeficiency virus
* Active infection requiring therapy, positive tests for hepatitis B surface antigen or hepatitis C ribonucleic acid (RNA)
* Active autoimmune disease, history of autoimmune disease or history of syndrome that required systemic steroids or immunosuppressive medications, e.g. organ, tissue, or allogenic hematopoietic stem cell transplant (HSCT) recipients. Exceptions include those with vitiligo or resolved childhood asthma/atopy. Subjects with asthma who require intermittent use of bronchodilators (such as albuterol) will not be excluded from this study
* Use of any live vaccines against infectious diseases up to 4 weeks (28 days) before receiving nivolumab. (NOTE: Inactivated seasonal influenza vaccines are permitted and do not require a 4-week waiting period before starting study treatment).
* Prisoners or subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness
* Patients with both brain and spine metastases will be excluded from the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse events (SAE) graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) version 4.0 | Up 12 weeks after first dose of study treatment
  All SAEs will be tabulated by type and grade. Proportion of individual type of SAE event will be estimated using the binomial distribution along with 95% confidence interval (exact method).

SECONDARY OUTCOMES:
Changes in the immune profile of peripheral blood during and after treatment with nivolumab in combination with stereotactic radiosurgery (immune response) | Baseline to up to 12 months
  Correlative outcomes will be summarized using descriptive statistics. Logistic regression model will be considered to explore potential association between the control rate and correlative outcomes.
Incidence of toxicity graded according to the NCI CTC 4.0 | Up to 30 days after completion of study treatment
  Toxicity events will be tabulated by type and grade. The severity and frequency of the toxicity will be tabulated by the tested dose or doses using descriptive statistics. The proportions of patient who experienced grade 3 or above toxicities will be estimated, along with 95% confidence intervals by each type of toxicity.
Local control rate in brain defined as no change in number of lesions at initial treatment in the brain and change on size of targeted lesion is =< 25% from initial measurement | From date of initial nivolumab treatment to first date that progressive disease is objectively documented, assessed up to 3 years
  The local control rate will be estimated using binomial distribution along with 95% confidence. The duration of the local control will be summarized using median and range.
Progression-free survival according to Response Evaluation Criteria in Solid Tumors criteria 1.1 | From the date of initial diagnosis (at surgery) to the date of progressive disease was defined (documented), assessed up to 3 years
  The probability of progression-free survival will be estimated using the Kaplan-Meier method.
Systematic control rate in spine defined as no change in number of lesions at initial treatment in the spine and change on size of targeted lesion is =< 25% from initial measurement | Up to 3 years
  The systematic control rate will be estimated using binomial distribution along with 95% confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Kleinberg, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (1):
- Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland, United States